CLINICAL TRIAL: NCT04811703
Title: Phase I Dose Escalation Study Evaluating the Safety of Adding Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) With Cisplatin-doxorubicin to the Systemic Chemotherapy, and the Recommended Phase II Dose, in Women With Insufficient Response to Carboplatin-paclitaxel for Advanced Epithelial Cancer of the Ovary, Fallopian Tubes or Peritoneum
Brief Title: Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Associated With Systemic Chemotherapy in Women With Advanced Ovarian Cancer
Acronym: PIPACOVA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL20_0920
Record Dates: First submitted 2021-03-08; First posted 2021-03-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Ovarian Carcinoma; Peritoneal Carcinomatosis; Stage III Ovarian Cancer; Stage IV Ovarian Cancer; Stage III Fallopian Tube Cancer; Stage IV Fallopian Tube Cancer; Metastatic Malignant Neoplasm in the Peritoneum
Keywords: Dose escalation; Phase I study; Intravenous Chemotherapy; Intraperitoneal chemotherapy; PIPAC; RP2D; cytoreductive surgery; Ovarian epithelial cancer; peritoneal cancer; doxorubicin; cisplatin; CA-125 antigen; pharmacokinetic
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined PIPAC / IV chemotherapy treatment (Experimental): Patients will undergo 3 cycles of combined chemotherapy, consisting of PIPAC (cisplatin-doxorubicin, escalating doses) and systemic chemotherapy (paclitaxel-carboplatine, standard doses). First patient will be treated at the lowest dose: doxorubicin 2.1 mg/m² and cisplatin 10.5 mg/m². Subsequent patients will be treated at the dose recommended by the CRM algorithm in the absence of dose-limiting toxicity. A total of 11 dose levels with a factor between 1 and 3 are considered. The maximum dose considered will be doxorubicin, 6.3 mg/m² and cisplatin, 31.5 mg/m². The doses of intravenous chemotherapy will be defined in a standard way, according to the habits of the investigating clinicians and in accordance with the doses received previously. Each cycle will last 28 days and will begin at day 1 with PIPAC procedure and will be completed at day 8 with systemic chemotherapy. Combined chemotherapy will be repeated every 4 weeks for up to 3 cycles in the absence of unacceptable toxicity.
  Interventions: Drug: Combined PIPAC / IV chemotherapy treatment

INTERVENTIONS:
Drug: Combined PIPAC / IV chemotherapy treatment — Addition of cisplatin-doxorubicin PIPAC sessions to carboplatin-paclitaxel systemic Chemotherapy

SUMMARY:
Women with history of tumor response insufficient to allow complete cytoreductive surgery after three cycles of previous neoadjuvant systemic carboplatin-paclitaxel chemotherapy will be prospectively recruited in this trial. After signed consent and if unresectability is confirmed, patients will undergo three cycles of doxorubicin-cisplatin PIPAC chemotherapy associated with systemic carboplatin-paclitaxel chemotherapy (alternating PIPAC and intravenous chemotherapy sessions over 3 cycles of 4 weeks).

The primary objective of the study is to determine the maximum tolerated dose (MDT).

During cycle 1, limiting dose toxicity must be collected as soon as it is known. Each patients will be treated at the dose recommended by the CRM (Continual Reassessment Method ) algorithm conditional on dose-limiting toxicity during Cycle 1.

The dose escalation will be guided by CRM to determine the recommended dose of PIPAC chemotherapy for phase II trial.

Secondary objectives are :

* to evaluate the anatomopathological response, the radiologic tumoral response and the evolution of the peritoneal cancer extent, to the combined chemotherapy
* to describe the pharmacokinetic of the PIPAC chemotherapy
* to investigate the KELIM parameter as a predictive marker in the response sensitivity of the combined chemotherapy treatment
* and to evaluate the safety of the combined chemotherapy. During the first day of the first cycle, blood samples will be collected to measure doxorubicin and cisplatin (pharmacokinetic study). Along these 3 cycles, the dose of antigen CA-125 will be performed before each chemotherapies (intraperitoneal or intravenous).

At the end of combined chemotherapy treatment, patients will undergo radiologic tumoral response by imaging assessment (scanner or MRI) and a last dosage of CA-125 will be realized..

In case of a complete / partial response / stabilization (RECIST criteria v.1.) on the imaging, re-evaluation for resectability will be done. If resectable disease, cytoreductive surgery will be programmed and a post-operative visit 1 month later will be realized. Otherwise for patients with progress disease or unresectable the participation in the study will be finished.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤ 75 years
* ECOG PS 0-2 ;
* Epithelial stage IIb to IVa carcinoma of the ovary, fallopian tubes, or peritoneum proven histologically, stage III or IV of the FIGO classification and with history of insufficient tumor response/ after three cycles of previous neoadjuvant systemic carboplatin-paclitaxel chemotherapy as judged by the investigators after discussion and validation in Multidisciplinary Team ;
* Adequate hematologic function
* Absolute Neutrophil Count > 1500 / mm3 (or 1.5 10 9/L)
* Hemoglobin ≥ 9.0 g/dL,
* platelets > 100 G/L,
* Adequate hepatic and renal function:
* Serum creatinine ≤1.5 times upper normal values or glomerular filtration rate ≥ 60 mL/min/1.73 m2 estimated by the CKD-EPI equation
* Total bilirubin ≤1.5 times the upper normal limit,
* ASAT / ALAT ≤1.5 times the upper normal limit (≤5 times upper normal limits for patients with liver metastases);
* Absence of unstable pathologies : myocardial infarction within 6 months prior to the start of the study, congestive heart failure, unstable angina, active cardiomyopathy, unstable rhythm disorder, uncontrolled hypertension, uncontrolled psychiatric disorders, severe infection, peptic ulcer, or any pathology that could be aggravated by treatment or limit compliance (investigator's judgment)
* Patient information given and Written informed consent obtained prior to the initiation of any specific study procedure
* Affiliated to a social insurance regime or similar

Exclusion Criteria:

* Extra-peritoneal metastases (position or number which make the disease unresectable)
* Signs of intestinal obstruction or lesions with risk of intestinal perforation, or signs of inflammatory disease of the digestive tract
* Contraindication to systemic chemotherapy CARBOPLATIN-PACLITAXEL :known allergy to paclitaxel
* Contraindication to the PIPAC procedure:
* Known allergy to cisplatin or other platinum-containing compounds
* Known allergy to doxorubicin or other anthracyclines or anthracenediones;
* Heart failure with myocardial insufficiency
* Uncontrolled coronary insufficiency;
* Pregnancy or breastfeeding
* Persons deprived of liberty or under guardianship ;
* Major patient protected by the Law;
* Persons participating in other research with an exclusion period still in progress at the time of inclusion or research that may interfere with the results of the present study (investigator's judgment) ;
* Impossibility to submit to the medical follow-up of the trial for geographical, social or psychic reasons (investigator's judgement)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities | First cycle of combined chemotherapy = day 1 up to day 28 of the first cycle
  Dose-limiting toxicities will be defined as any of the following events observed during the first cycle of treatment and judged by the investigator to be possibly related to the treatment, based on the classification of the National Cancer Institute Common Criteria for Adverse Events Terminology (NCI CTCAE) Version 5.0 :
  * Grade 4 Neutropenia (absolute neutrophil count <500 /mm3 (or 0.5 109/L)) ≥7 consecutive days;
  * Neutropenia of grade ≥ 3 (absolute neutrophil count <1000 /mm3 (or 1 109/L)) and temperature ≥ 38.5°C ;
  * Thrombocytopenia grade 4 (<25,000/mm3 platelets (or 25 109/L)) or grade 3 (< 50,000/mm3 (or 50 109/L)) associated with bleeding ;
  * Non-hematological toxicity of grade ≥3 (excluding non-life-threatening toxicities such as alopecia, asymptomatic hypophosphatemia, etc.) despite adequate medical intervention judged by the investigator

SECONDARY OUTCOMES:
Rate of complete surgical resection | During cytoreductive surgery performed at the end of cycle 3 of combined chemotherapy (each cycle is 28 days), and at a maximum of 12 weeks after the third cycle of PIPAC
  Assessed during cytoreductive surgery by the Completeness Cytoreduction (CC) score after the 3 cycles of combined chemotherapy.
  Complete cytoreduction refers to a CC-0 or CC-1 score whereas a CC-2 or 3 score is classified as incomplete ; CC-0 score indicates no evidence of macroscopic disease after cytoreduction, a CC-1 score indicates persisting microscopic disease (tumour nodules are < 2.5 mm), a CC-2 score indicates persisting macroscopic disease (residual tumour nodules between 2.5 mm and 2.5 cm) and finally a CC-3 score indicates tumour nodules > 2.5 cm or a confluence of unresected tumour.
Proportion of complete, partial or stabilized tumor response | After completing chemotherapy treatment, at 4 to 5 weeks after the third cycle of post PIPAC (each cycle is 28 days)
  Assessed according to the Response Evaluation Criteria in Solid Tumor (RECIST) criteria version 1.1, on thoracic abdominal pelvic imaging (scanner or MRI in case of contraindication).
Peritoneal cancer index (PCI) evolution | At day 1 of the beginning of each cycle during PIPAC procedure, at 4 to 5 weeks post PIPAC cycle 3 (each cycle is 28 days) and during post-treatment laparoscopy and/or during cytoreductive surgery (12 weeks max post PIPAC cycle 3)]
  PCI index will be evaluated under videosurveillance during laparoscopy. PCI is determined according to Sugarbaker, based on lesion size and distribution. Using a pictorial of the abdomen, each location of a 13 point list receives a peritoneal cancer grade ranging from 0 to 3. The counts for all 13 locations are then summarized as PCI.
Area under the curve (AUC) for plasma concentration of DOXORUBICIN and CISPLATIN | During day 1 of the first cycle of PIPAC chemotherapy (at 0, 30 minute, 1 hour, 2 hours, 4 hours, 6 hours, 7/8 hours and 24 hours post PIPAC for the both chemotherapeutic compound and 48 hours only for DOXORUBICIN), each cycle being 28 days.
  The plasma biodisponibility of the PIPAC doxorubicin and CISPLATIN (total and ultrafilterable platinum) chemotherapeutic compound will be assessed by reporting the Area under the plasma concentration- time curve.
Change in CA-125 concentration | Pharmacokinetic blood samples for each cycle, each cycle being 28 days (at day 1 for PIPAC chemotherapy; at day 8 for systemic chemotherapy) and before post-treatment laparoscopy at 4-5 weeks after the third PIPAC)
  CA-125 evolution profile will be monitored during chemotherapy and before surgery of reevaluation at post-treatment visit. Then, mathematical modeling of CA-125 elimination rate KELIM will be calculated from individual CA-125 levels.
Rates of adverse events and operative complications | Up to 8 months after inclusion
  Adverse events according to the NCI CTCAE v5.0 classification (including toxicities) and per- and post-operative complications according to the Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Justine ARQUILLIERE, MD, Principal Investigator — Hospices Civils de Lyon
Locations (6):
- France (6):
  - Hôpital Claude Huriez - Chirurgie générale et digestive, Lille
  - Hôpital Claude Huriez - Oncologie médicale, Lille
  - Hôpital de la Croix-Rousse, Lyon
  - Hôpital Lyon Sud - Chirurgie Digestive et Oncologique, Pierre-Bénite
  - Hôpital Lyon Sud - Chirurgie Gynécologique et oncologique-obstétrique, Pierre-Bénite
  - Hôpital Lyon Sud - Oncologie Médicale, Pierre-Bénite